CLINICAL TRIAL: NCT06062758
Title: The Effect of Simulation-Based Electroconvulsive Therapy Training on Perception and Knowledge of Nursing Students: A Semi-Experimental Study
Brief Title: The Efficiency of Simulation-Based Electroconvulsive Therapy Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fenerbahce University (Other)
Collaborators: New York University (Other)
Responsible Party: Principal Investigator, Gül DİKEÇ, Assoc. Prof., Fenerbahce University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Fenerbahce University
Record Dates: First submitted 2023-09-14; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: ECT; Mental Disorder; Nursing Caries
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Simulation training will consist of three stages. The first stage is preliminary preparation. At this stage, students who review the resources identified and come prepared for the simulation scenario will be asked questions appropriate to the simulation objectives to help them remember the subject. In the second stage, the simulation will be realized. A high-fidelity mannequin/simulator will be used during the simulation, and the responsible faculty will give patient responses in the cabin. While the students taking roles during the simulation provide care to the patient, other group members will watch their teammates in the cabin or in a The simulation will be finalized by discussing the critical points of the case, the care to be given, communication skills and patient safety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nursing Students (Experimental): The study population will consist of fourth-year students (n=72) of Fenerbahçe University Faculty of Health Sciences, Department of Nursing, Turkish Nursing Program. Sampling calculation and sample selection will not be made in the study, aiming to reach the entire population.
  Interventions: Behavioral: ECT Simulation Training

INTERVENTIONS:
Behavioral: ECT Simulation Training — Simulation training will consist of three stages. The first stage is preliminary preparation. At this stage, students who review the resources identified and come prepared for the simulation scenario will be asked questions appropriate to the simulation objectives to help them remember the subject. In the second stage, the simulation will be realized. A high-fidelity mannequin/simulator will be used during the simulation, and the responsible faculty will give patient responses in the cabin. While the students taking roles during the simulation provide care to the patient, other group members will watch their teammates in the cabin or in a The simulation will be finalized by discussing the critical points of the case, the care to be given, communication skills and patient safety.

SUMMARY:
The goal of this study is to determine the effect of the simulation-based Electroconvulsive Therapy (ECT) Simulation Training applied to senior nursing students studying at a foundation university on students' perceptions and knowledge levels about ECT.

The research hypotheses are as follows; H0: There is no significant difference between students' perception and knowledge levels about ECT before and after simulation-based ECT training to be applied to nursing students.

H1: There is a significant difference between students' perception and knowledge levels about ECT before and after the simulation-based ECT training to be applied to nursing students.

Type of study: This study was planned in a single group pre-test post-test quasi-experimental design.

Participants: The study population will consist of fourth-year students (n=72) of Fenerbahçe University Faculty of Health Sciences, Department of Nursing, Turkish Nursing Program.

Intervention: The study will collect data before the students start clinical practice and before the theoretical course on Electroconvulsive Therapy. Then, a one-hour theoretical training on electroconvulsive therapy will be given. This training includes ECT, its history, use areas, nursing care before, during and after ECT and patient education. After the theoretical lecture, a simulation scenario will be distributed to the students, and they will be asked to come prepared on the simulation day. Students will be divided into groups of 15 people, and the groups will be met in the Simulation Laboratory at the determined group hours.

Control Group: There is no control group. Outcome: Perceptions and knowledge levels about ECT.

DETAILED DESCRIPTION:
Aim This study aimed to determine the effect of the simulation-based Electroconvulsive Therapy Simulation Training applied to senior nursing students studying at a foundation university on students' perceptions and knowledge levels about ECT.

Study Design This study was planned in a single group pre-test post-test quasi-experimental design.

Hypotheses The research hypotheses are as follows; H0: There is no significant difference between students' perception and knowledge levels about ECT before and after simulation-based ECT training to be applied to nursing students.

H1: There is a significant difference between students' perception and knowledge levels about ECT before and after the simulation-based ECT training to be applied to nursing students.

Varıables Of The Study The study's dependent variable is the level of perception and knowledge about ECT, and the independent variable is ECT simulation training.

Settings The research is aimed to be implemented between 01.10.2023 05.01.2024 between 01.10.2023-and 01.01.2024 within the scope of the Psychiatric and Mental Health Nursing course and in the Simulation Laboratory of Fenerbahçe University, Faculty of Health Sciences, Department of Nursing, Turkish Nursing Program senior students.

Participants The study population will consist of fourth-year students (n=72) of Fenerbahçe University Faculty of Health Sciences, Department of Nursing, Turkish Nursing Program. Sampling calculation and sample selection will not be made in the study, aiming to reach the entire population.

Inclusion Criteria:

* Being a fourth-year student of Fenerbahçe University Faculty of Health Sciences, Department of Nursing, Turkish Nursing Program,
* To be enrolled in Mental Health and Diseases course,
* Volunteering to participate in the study.

Exclusion Criteria:

* Being a student of Fenerbahçe University, Faculty of Health Sciences, Department of Nursing, Turkish Nursing Program, but not enrolled in the Mental Health and Diseases course,
* Not participating in simulation training,
* Incomplete completion of data collection tools,
* Not volunteering to participate in the study. Measurements Data will be collected with the Information Form and the Perception and Knowledge Scale about ECT.

Information Form: The researcher prepared this form, consisting of questions about the students' sociodemographic characteristics and their familiarity with mental disorders and ECT.

Perception and Knowledge Scale about ECT: It was developed by Tsai et al. to determine knowledge and attitudes about ECT. It consists of 18 items in total. The subscale for perceptions about electroconvulsive therapy includes six items on a five-point Likert scale scored between 1 (strongly disagree) and 5 (strongly agree), and the subscale for knowledge about ECT includes 12 yes-no items. Total scale score changes between 12 and 60. Higher perception and knowledge subscale scores mean a better perception and higher level of knowledge. The Turkish validity and reliability of the scale was performed by Yıldırım et al. (2023). The Cronbach's alpha coefficient was 0.85 for the perception subscale and 0.78 for the knowledge subscale. Permission to use the scale was obtained from Dr. Yıldırım via e-mail.

Data Collection The study will collect data before the students start clinical practice and before the theoretical course on Electroconvulsive therapy. Then, a one-hour theoretical training on electroconvulsive therapy will be given. This training includes ECT, its history, use areas, nursing care before, during, and after ECT, and patient education. After the theoretical lecture, a simulation scenario will be distributed to the students, and they will be asked to come prepared on the simulation day. Students will be divided into groups of 15 people, and the groups will be met in the Simulation Laboratory at the determined group hours.

The coding method will match the students' pre-test, post-test, and follow-up scores. Students will be asked to code the codes consisting of the first letter of their surname, the last two digits of their date of birth, and their lucky numbers on the first page of the pre-test. They will be asked to repeat this coding in the post-test and follow-up.

The pre-test will apply the information Form and Perception and Knowledge Scale about ECT. Then, theoretical training and simulation training will be applied. Students will be asked to fill in the Perception and Knowledge Scale about ECT in the post-test (after two weeks of pre-test). Finally, a follow-up test will be conducted after the students complete the mental health and diseases nursing course and clinical practice (after three months later pre-test).

ECT Simulation Training ECT Simulation training prepared by the researcher consists of instructor and student scenarios. The faculty member scenario includes simulation learning objectives, detailed information about the case, possible facilitating patient and student questions and answers during the simulation, and an evaluation form. The student scenario includes simulation objectives, information about the case and roles, and an evaluation form.

Simulation training will consist of three stages. The first stage is preliminary preparation. At this stage, students who review the resources identified and come prepared for the simulation scenario will be asked questions appropriate to the simulation objectives to help them remember the subject. Then, four students will be selected from the groups and given their roles. In the second stage, the simulation will be realized. A high-fidelity mannequin/simulator will be used during the simulation, and the responsible faculty member and researcher will give patient responses in the cabin. While the students taking roles during the simulation provide care to the patient, other group members will watch their teammates in the cabin or in a classroom where a camera is provided. The third stage is the debriefing stage. At this stage, three evaluations will be made. First, the self-evaluation of the students who took part in the simulation, then the evaluation of the students by their groupmates, and finally, the evaluation of the faculty member will be shared. The simulation will be finalized by discussing the critical points of the case, the care to be given, communication skills and patient safety.

Data Analysis The data obtained in the study will be analyzed using SPSS (Statistical Package for Social Sciences) for the Windows 26.0 program. The data will be analyzed by number, percentage distributions, mean and standard deviation. Kurtosis and Skewness will be used to evaluate whether the scale scores are normally distributed, and paired t-tests or Wilcoxon signed-rank tests will be used to compare the pre-test and post-test scores. All data will be tested for significance at p<0.05 level.

Funding No expenditure will be made on any item other than the consumables of the existing forms for the research. The researcher will cover stationery and consumables.

In addition, the simulator (high fidelity mannequin) in the simulation laboratory of Fenerbahçe University Faculty of Health Sciences, Department of Nursing will be used within the scope of the study by obtaining the necessary permissions.

ELIGIBILITY:
Inclusion Criteria:

* Being a fourth-year student of Fenerbahçe University Faculty of Health Sciences, Department of Nursing, Turkish Nursing Program,
* To be enrolled in Psychiatric and Mental Health course,
* Volunteering to participate in the study.

Exclusion Criteria:

* Being a student of Fenerbahçe University, Faculty of Health Sciences, Department of Nursing, Turkish Nursing Program, but not enrolled in the Mental Health and Diseases course,
* Not participating in simulation training,
* Incomplete completion of data collection tools,
* Not volunteering to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-10-02 (Estimated); Primary Completion 2023-10-18 (Estimated); Study Completion 2024-01-03 (Estimated)

PRIMARY OUTCOMES:
Perception and Knowledge about ECT | Pre-test (before the intervention), post-test (two weeks after intervention) and three months after follow up
  Perception and Knowledge Scale about ECT

CONTACTS AND LOCATIONS:
Locations (1):
- Fenerbahce University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The coding method will match the students' pre-test, post-test and follow-up scores. Students will be asked to code the codes consisting of the first letter of their surname, the last two digits of their date of birth, and their lucky numbers on the first page of the pre-test. They will be asked to repeat this coding in the post-test and follow-up.

REFERENCES:
- [Derived] Dikec G, San EO. The Effect of Simulation-Based Electroconvulsive Therapy Education on Perception and Knowledge of Nursing Students: A Semiexperimental Study. J ECT. 2025 Feb 25. doi: 10.1097/YCT.0000000000001130. Online ahead of print. PMID 40020048